CLINICAL TRIAL: NCT06526078
Title: A Brief Automated Neurocognitive Training to Enhance the Real-World Impact of Ketamine's Rapid Antidepressant Effect
Brief Title: Cognitive Training as an Adjunct to Ketamine in Real-world Clinics
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rebecca Price, Associate Professor of Psychiatry and Psychology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY23110120; R01MH136179 (NIH); R01MH136178 (NIH)
Record Dates: First submitted 2024-07-22; First posted 2024-07-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Training (Experimental): Web-based cognitive training
  Interventions: Behavioral: Cognitive Training
- Sham Training (Sham Comparator): Web-based sham training
  Interventions: Behavioral: Sham Training

INTERVENTIONS:
Behavioral: Cognitive Training — Sessions of cognitive training exercises (15-20min each) self-administered via a web app
  Arms: Cognitive Training
Behavioral: Sham Training — Sessions of sham training exercises (15-20min each) self-administered via a web app
  Arms: Sham Training

SUMMARY:
In a sample of patients already receiving ketamine (or esketamine) treatment as part of their clinical care, this project seeks to test whether we can enhance and/or extend (es)ketamine's rapid effects by introducing helpful information delivered by a computer-based cognitive training protocol. This work could ultimately lead to the ability to treat depression more efficiently and with broader dissemination by rapidly priming the brain for helpful forms of learning.

ELIGIBILITY:
Inclusion Criteria:

1. be between the ages of 18 and 80 years
2. score ≥20 on the Montgomery-Asberg Depression Rating Scale (MADRS)
3. per SCID-5-RV interview, meet DSM-5 diagnostic criteria for at least one of the following: Major Depressive Disorder, Bipolar Disorder (I or II), Persistent Depressive Disorder, or Other Specified Depressive or Bipolar Disorder
4. exhibit treatment resistance, defined as: (a) failure to respond to ≥1 adequate trials of an evidence-based treatment for mood disorder [per the Antidepressant Treatment History Form-Short Form Modified Score Sheet (ATHF-SF-Modified)] and/or (b) failure to respond to ≥1 adequate mood stabilizer or other evidence-based treatment trials (for bipolar depression patients) and/or (c) a history of intolerance during attempted trials of evidence-based treatments for mood disorders and/or (d) failure to respond to ≥1 prior treatment trials (e.g., medication, psychotherapy) for Post Traumatic Stress Disorder (PTSD)
5. be eligible and clinically enrolled for an upcoming ketamine or esketamine induction series at one of our study clinics according to that clinic's standard intake procedures
6. agree to maintain a stable schedule of concomitant psychiatric medications throughout the ketamine induction phase (minor adjustments to PRN meds and timing of meds are allowable), and for 4 weeks post-induction phase
7. possess a level of judgment and understanding sufficient to agree to all procedures required by the protocol and must sign an informed consent document
8. be willing and able to provide names and contact information for at least 1 additional emergency contact in the patient's proximal geographic area (in addition to the ketamine treatment team at the enrolling site)

Exclusion Criteria:

1. Presence of current/acute psychosis, mania, or dementia, or a diagnosis of developmental disorder with significant language and/or intellectual impairment (e.g., autism spectrum disorder)
2. Current/acute suicide risk with intent to act, defined as CSSRS past-week ideation score ≥ 4 among outpatients; patients engaged in residential or inpatient care at the time of enrollment need not meet this CSSRS score criterion, as their current/acute suicide risk is extremely low by virtue of the residential/inpatient, round-the-clock care they are already receiving at time of enrollment
3. Concern for dementia or significant cognitive decline, per interviewer observations and impressions during screening assessments
4. Current pregnancy or breastfeeding
5. English reading level <5th grade as per patient self-report Rationale: to ensure adequate reading comprehension for verbal ASAT/sham stimuli which are presented in English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale: During (Es)Ketamine Induction | Trajectories from baseline through end of 'induction phase' treatments (up to max of 12 weeks)
  depression severity; range 0-60; high score=worse outcome
Montgomery Asberg Depression Rating Scale: After (Es)Ketamine Induction | Trajectories from final 'induction phase' treatment through 4 weeks post-induction
  depression severity; range 0-60; high score=worse outcome

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptoms | Trajectories from baseline through 12 months post-induction
  Self-reported depression (range: 0-27; higher scores = worse outcome)
PROMIS Measures-depression | Trajectories from baseline through 12 months post-induction
  Patient-Reported Outcomes Measurement Information System (PROMIS) measure: Self-reported depression T-score range: 0-100 (higher score = worse outcome)
Beck Hopelessness Scale | Trajectories from baseline through 12 months post-induction
  self reported to measure key aspects of hopelessness; range = 0-20, higher score=worse outcome
PROMIS Measures-anxiety | Trajectories from baseline through 12 months post-induction
  Patient-Reported Outcomes Measurement Information System (PROMIS) measure: Self-reported anxiety T-score range: 0-100 (higher score = worse outcome)
PROMIS Measures-anger | Trajectories from baseline through 12 months post-induction
  Patient-Reported Outcomes Measurement Information System (PROMIS) measure: Self-reported anger T-score range: 0-100 (higher score = worse outcome)
PROMIS Measures-Positive Affect | Trajectories from baseline through 12 months post-induction
  Patient-Reported Outcomes Measurement Information System (PROMIS) measure: Self-reported positive affect/well-being T-score range: 0-100 (higher score = better outcome)
PROMIS Measures-Sleep Disturbance | Trajectories from baseline through 12 months post-induction
  Patient-Reported Outcomes Measurement Information System (PROMIS) measure: Self-reported sleep disturbance T-score range: 0-100 (higher score = worse outcome)
PROMIS Measures-Cognitive Function | Trajectories from baseline through 12 months post-induction
  Patient-Reported Outcomes Measurement Information System (PROMIS) measure: Self-reported cognitive function T-score range: 0-100 (higher score = better outcome)
Cognitive Triad Inventory | Trajectories from baseline through 12 months post-induction
  Negative perceptions of self, future, & world (range=36-252; higher score = better outcome)
Montgomery Asberg Depression Rating Scale: Naturalistic Follow-up | Trajectories from baseline through 12 months post-induction
  depression severity; range 0-60; high score=worse outcome

OTHER OUTCOMES:
Implicit Association Test | Trajectories from baseline through 4 weeks post-induction
  performance-based "target engagement" measure of implicit self-esteem; range = -inf-inf; high score=worse outcome
Columbia Suicide Severity Rating Scale--Intensity of Most Severe Ideation | Trajectories from baseline through 12 months post-induction
  suicidal ideation/thoughts; range 0-5; high score=worse outcome
Patient Health Care Utilization Survey (PHCUS) | Trajectories from baseline through 12 months post-induction
  interview measure of psychiatric and healthcare service utilization
PROMIS Measures-substance Use | Trajectories from baseline through 12 months post-induction
  Patient-Reported Outcomes Measurement Information System (PROMIS) measure: Self-reported substance use Raw score range: 0-35 (higher score = worse outcome)
PROMIS Measures-alcohol | Trajectories from baseline through 12 months post-induction
  Patient-Reported Outcomes Measurement Information System (PROMIS) measure: Self-reported alcohol use T-score range: 0-100 (higher score = worse outcome)
Acceptability, Appropriateness, and Feasibility | Post-Induction Week 1 assessment (approximately 1-7 days post induction)
  self-report scales of intervention acceptability, appropriateness, feasibility; range = 5-20; high score=better rating
Short Form Health Survey | Baseline through 12 months post-induction
  Self-report measure of Quality-Adjusted Life-Years (QALYs)
Client Satisfaction Questionnaire (CSQ-8) | Post-Induction Week 1 assessment (approximately 1-7 days post induction)
  Self-reported satisfaction; range: 8-32; high score=better rating
mHealth App Usability Questionnaire (MAUQ) | Post-Induction Week 1 assessment (approximately 1-7 days post induction)
  Self-reported usability of cognitive training web app; range = 18-126; high score=better rating
Qualitative interviews assessing implementation | 12 months post-induction
  Custom qualitative interviews with qualitative coding
Compliance with prescribed cognitive training sessions | Throughout the entirety of three discrete CT "bursts"
  Compliance data from web app logs
PROMIS Measures-Social Functioning | Trajectories from baseline through 12 months post-induction
  Patient-Reported Outcomes Measurement Information System (PROMIS) measures of social functioning: T-score range: 0-100 (higher score = better outcome)
PROMIS Measures-Pain | Trajectories from baseline through 12 months post-induction
  Patient-Reported Outcomes Measurement Information System (PROMIS) measures of pain: T-score range: 0-100 (higher score = better outcome)
Awe Experience Scale (AWE-S) | 1 week after first induction treatment
  self-report measure of awe-inspiring experiences (range: 30-210; higher score=greater awe)
Implicit Association Test across follow-up | Trajectories through 12 months post-induction
  performance-based "target engagement" measure of implicit self-esteem; range = -inf-inf; high score=worse outcome
Time to relapse | Baseline through 12 months post-induction
  Time-to-event for relapse to within 25% of baseline MADRS score
Time to first maintenance treatment | Baseline through 12 months post-induction
  Time-to-event for the date of return to clinic for first maintenance treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca B Price, PhD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - Kaiser Foundation Research Institute, a division of Kaiser Foundation Hospitals, Oakland, California
  - University of Illinois at Chicago, Chicago, Illinois
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results will be shared with other researchers via the NIMH Data Archive (NDA) data repository.
Time Frame: Data will become available one year after study completion and will be available indefinitely.
Access Criteria: NDA access required.
URL: https://nda.nih.gov/